CLINICAL TRIAL: NCT03437304
Title: A Phase I/II, Randomised, Multicentre, Placebo-controlled, Partially-blinded, Parallel-group Study to Assess the Safety, Tolerability and Immune Response Following Vaccination With Immunose™ FLU in Older Adults (Age 50 to 75 Years)
Brief Title: Study to Assess the Safety, Tolerability and Immune Response Following Vaccination With Immunose™ FLU in Older Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eurocine Vaccines AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EURO 17-09
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Influenza
Keywords: Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Immunose™ FLU 1% (Experimental): Immunose™ FLU 1%. QIV, 30 μg HA/strain and 1% Endocine™ 200 μl for intranasal administration, 2 dosing occasions.
  Interventions: Biological: Immunose™ FLU 1%
- Immunose™ FLU 2%, 200 μl (Experimental): Immunose™ FLU 2%. QIV, 30 μg HA/strain and 2% Endocine™, 200 μl for intranasal administration, 2 dosing occasions.
  Interventions: Biological: Immunose™ FLU 2%, 200 μl
- Immunose™ FLU 2%, 300 μl (Experimental): Immunose™ FLU 2%, 300 μl. QIV, 30 μg HA/strain and 2% Endocine™, 300 μl for intranasal administration, 2 dosing occasions.
  Interventions: Biological: Immunose™ FLU 2%, 300 μl
- Influenza antigen (Experimental): Influenza antigen. QIV, 30 μg HA/strain, 200 μl for intranasal administrations, 2 dosing occasions.
  Interventions: Biological: Influenza antigen
- Placebo (Placebo Comparator): Placebo. Saline (NaCl), 200 μl for intranasal administration, 2 dosing occasions.
  Interventions: Drug: Placebo
- i.m comparator and Immunose™ FLU 2% (Experimental): i.m comparator: QIV 15 μg HA/strain, 500 µl for a single intramuscular administration, and Immunose FLU 2%: QIV 30 μg HA/strain and 2% Endocine™, 200 μl for intranasal administration. A second dose of Immunose FLU 2% will be administered 3 weeks later.
  Interventions: Biological: Immunose™ FLU 2%, 200 μl; Biological: i.m comparator
- i.m comparator (Active Comparator): i.m comparator. QIV 15 μg HA/strain, 500 µl for a single intramuscular administration.
  Interventions: Biological: i.m comparator

INTERVENTIONS:
Biological: Immunose™ FLU 1% — Quadrivalent influenza vaccine with 30 μg HA/strain and 1% Endocine™, dosing volume 200 μl, intranasal administration x 2
  Arms: Immunose™ FLU 1%
Biological: Immunose™ FLU 2%, 200 μl — Quadrivalent influenza vaccine with 30 μg HA/strain and 2% Endocine™, dosing volume 200 μl, intranasal administration x 2
  Arms: Immunose™ FLU 2%, 200 μl; i.m comparator and Immunose™ FLU 2%
Biological: Immunose™ FLU 2%, 300 μl — Quadrivalent influenza vaccine with 30 μg HA/strain and 2% Endocine™, dosing volume 300 μl, intranasal administration x 2
  Arms: Immunose™ FLU 2%, 300 μl
Biological: Influenza antigen — Quadrivalent influenza vaccine with 30 μg HA/strain, dosing volume 200 μl, intranasal administration x 2
  Arms: Influenza antigen
Drug: Placebo — NaCl dosing volume 200 μl, intranasal administration x 2
  Other Names: Saline (NaCl)
  Arms: Placebo
Biological: i.m comparator — Quadrivalent influenza vaccine containing 15 μg HA/strain, 500 µl for intramuscular administration x 1
  Arms: i.m comparator; i.m comparator and Immunose™ FLU 2%

SUMMARY:
This is a Phase I/II, randomised, multicentre, partially double-blind (group 1, 2, 4 and 5), parallel-group study designed to primarily evaluate the safety, tolerability and immune response in older adults (age 50 to 75 years) following Immunose™ FLU vaccination at 5 sites in Sweden. A total of 300 subjects will be randomised to 1 of 7 treatment groups. The hypothesis is that Immunose™ FLU is safe and tolerable and will increase the influenza-specific mucosal immune response in older adults.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study related procedures.
2. Male or female 50 to75 years of age (both inclusive) at screening.
3. Subjects who the Investigator believes will comply with the requirements of the protocol.
4. Judged by the Investigator to have no serious illness based on medical history, physical examination, ECG, vital signs and blood and urine assessments at screening.
5. All females should have been post-menopausal for at least 12 months or use a highly effective contraceptive method to prevent pregnancy. Non-menopausal females have to use contraceptive methods with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen- only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD], intrauterine hormone-releasing system [IUS], bilateral tubal occlusion, sexual abstinence). Any male partner should be willing to use condom or should be vasectomized.

Exclusion Criteria:

1. Diagnosis of laboratory-confirmed influenza in the 2017/2018 season.
2. Use of any investigational drug product within 3 months before screening or planned use during the study period, including the safety follow-up period.
3. Administration of an influenza vaccine during the 9 months before screening.
4. Previously received another vaccine within 28 days before administration of the study vaccine, or is scheduled to receive another vaccine during the study period, excluding the safety follow-up period.
5. Any contra-indication to intramuscular administration of the comparator influenza vaccine according to its SPC.
6. History of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study vaccine (e.g., to eggs or egg product as well as ovalbumin, chicken protein, chicken feathers, influenza viral protein, kanamycin, gentamycin, neomycin sulphate, formaldehyde and sodium deoxycholate).
7. Diagnosis of asthma with poor disease control as assessed by the Investigator.
8. Potent immunosuppressive therapy including cytostatics, antibodies, drugs acting on immunophilins, interferons and other drugs used to prevent rejection of organ transplants, within 6 months before screening.
9. Use of any parenteral or oral corticosteroids within 30 days prior to screening. Inhaled steroids are allowed.
10. Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
11. Any progressive or severe neurologic disorder, seizure disorder or Guillain-Barré syndrome.
12. Any history of Guillain-Barré syndrome.
13. Received blood, blood products and/or plasma derivatives or any administration of immunoglobulin preparation within the 3 months prior to Visit 2, or planned during the study.
14. Participation in blood donation within 3 months or plasma donation within 1 month prior to Visit 2.
15. History of substance or alcohol abuse within the past 2 years.
16. History or any illness/condition that, in the opinion of the Investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
17. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody or HIV.
18. Pregnant or lactating female or intent to become pregnant during the clinic phase and for 2 months after the last vaccination.
19. History of Bell's palsy.
20. Ongoing regular use of intranasal sprays including corticosteroids and decongestants.
21. Ongoing cough, sinusitis, allergic rhinitis, nasal polyps or obstruction, including septum deviation significant enough to prevent bilateral administration of study vaccine.
22. Known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
23. Subjects that are prone to nosebleed.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, during the clinical phase. | Visit 2 (Day 0)
  Type and incidence of AEs and SAEs. Treatment group 1-7.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, during the clinical phase. | Visit 3 (Day 21)
  Type and incidence of AEs and SAEs. Treatment group 1-7.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, during the clinical phase. | Visit 4 (Day 42)
  Type and incidence of AEs and SAEs. Treatment group 1-6.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, during the safety follow-up phase. | Day 90
  Type and incidence of AEs and SAEs of special intrerest. Treatment group 7.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, during the safety follow-up phase. | Day 111
  Type and incidence of AEs and SAEs of special intrerest. Treatment group 1-6.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, during the safety follow-up phase. | Day 180
  Type and incidence of AEs and SAEs of special intrerest. Treatment group 7.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, during the safety follow-up phase. | Day 201
  Type and incidence of AEs and SAEs of special intrerest. Treatment group 1-6.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, during the treatment visits. | Visit 2 (Day 0)
  Frequency and severity of discomfort in the nose and/or throat before study drug administration and at 15, 30, 60 and 120 minutes after study drug administration. Treatment group 1-5.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, during the treatment visits. | Visit 2 (Day 0)
  Frequency and severity of discomfort in the nose and/or throat and/or arm before study drug administration and at 15, 30, 60 and 120 minutes after study drug administration. Treatment group 6.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, during the treatment visits. | Visit 2 (Day 0)
  Frequency and severity of discomfort in the arm before study drug administration and at 15, 30, 60 and 120 minutes after study drug administration. Treatment group 7.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, during the treatment visits. | Visit 3 (Day 21)
  Frequency and severity of discomfort in the nose and/or throat before study drug administration and at 15, 30, 60 and 120 minutes after study drug administration. Treatment group 1-6.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, from baseline to last clinic visit. | Visit 1 (Day -42 to -1) to Visit 4 (Day 42)
  Frequency of clinically significant changes in ECG. Treatment group 1-6.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, from baseline to last clinic visit. | Visit 1 (Day -42 to -1) to Visit 3 (Day 21)
  Frequency of clinically significant changes in ECG. Treatment group 7.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, from baseline to last clinic visit. | Visit 1 (Day -42 to -1) to Visit 4 (Day 42)
  Frequency of clinically significant changes in vital signs. Treatment group 1-6.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, from baseline to last clinic visit. | Visit 1 (Day -42 to -1) to Visit 3 (Day 21)
  Frequency of clinically significant changes in vital signs. Treatment group 7.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, from baseline to last clinic visit. | Visit 1 (Day -42 to -1) to Visit 4 (Day 42)
  Frequency of clinically significant changes in physical examination findings. Treatment group 1-6.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, from baseline to last clinic visit. | Visit 1 (Day -42 to -1) to Visit 3 (Day 21)
  Frequency of clinically significant changes in physical examination findings. Treatment group 7.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, from baseline to last clinic visit. | Visit 1 (Day -42 to -1) to Visit 4 (Day 42)
  Frequency of clinically significant changes in laboratory variables. Treatment group 1-6.
Safety of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens, from baseline to last clinic visit. | Visit 1 (Day -42 to -1) to Visit 3 (Day 21)
  Frequency of clinically significant changes in laboratory variables. Treatment group 7.

SECONDARY OUTCOMES:
Evaluation of the immune response to Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens. | Visit 2 (Day 0)
  Measurement of HaemaggIutination-inhibition titers in serum. Treatment group 1-7.
Evaluation of the immune response to Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens. | Visit 3 (Day 21)
  Measurement of HaemaggIutination-inhibition titers in serum. Treatment group 1-7.
Evaluation of the immune response to Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens. | Visit 4 (Day 42)
  Measurement of HaemaggIutination-inhibition titers in serum. Treatment group 1-6.
Evaluation of the immune response to Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens. | Visit 2 (Day 0)
  Measurement of Virus Neutralization titers in serum. Treatment group 1-7.
Evaluation of the immune response to Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens. | Visit 3 (Day 21)
  Measurement of Virus Neutralization titers in serum. Treatment group 1-7.
Evaluation of the immune response to Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens. | Visit 4 (Day 42)
  Measurement of Virus Neutralization titers in serum. Treatment group 1-6.
Evaluation of the immune response to Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens. | Visit 2 (Day 0)
  Measurement of Single Radial Haemolysis titres in serum. Treatment group 1-7.
Evaluation of the immune response to Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens. | Visit 3 (Day 21)
  Measurement of Single Radial Haemolysis titres in serum. Treatment group 1-7.
Evaluation of the immune response to Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens. | Visit 4 (Day 42)
  Measurement of Single Radial Haemolysis titres in serum. Treatment group 1-6.
Evaluation of the immune response to Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens. | Visit 2 (Day 0)
  Measurement of Immunoglobulin A (IgA) titers in nasal secretion. Treatment group 1-7.
Evaluation of the immune response to Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens. | Visit 3 (Day 21)
  Measurement of Immunoglobulin A (IgA) titers in nasal secretion. Treatment group 1-7.
Evaluation of the immune response to Immunose™ FLU based on Endocine™ and quadrivalent influenza antigens. | Visit 4 (Day 42)
  Measurement of Immunoglobulin A (IgA) titers in nasal secretion. Treatment group 1-6.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rein Hedin, MD, Principal Investigator — CTC Clinical Trial Consultants AB
Locations (5):
- Sweden (5):
  - Site 5, Borås
  - Site 4, Helsingborg
  - Site 2, Linköping
  - Site 3, Malmo
  - Site 1, Uppsala

IPD SHARING:
Plan to Share IPD: No